CLINICAL TRIAL: NCT02399215
Title: Multicenter Phase 2 Study of Nintedanib for Patients With Advanced Carcinoid Tumors
Brief Title: Nintedanib in Treating Patients With Locally Advanced or Metastatic Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 259114; NCI-2015-00238 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 259114 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2015-03-13; First posted 2015-03-26 (Estimated); Results first posted 2022-06-28 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Carcinoid Tumor; Metastatic Carcinoid Tumor; Neuroendocrine Neoplasm
MeSH Terms: conditions — Carcinoid Tumor; Neuroendocrine Tumors | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (nintedanib) (Experimental): Patients receive nintedanib PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Nintedanib; Other: Pharmacological Study; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nintedanib — Given PO
  Other Names: BIBF 1120; BIBF-1120; Intedanib; Multitargeted Tyrosine Kinase Inhibitor BIBF 1120; tyrosine kinase inhibitor BIBF 1120; Vargatef
Other: Pharmacological Study — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies how well nintedanib works in treating patients with neuroendocrine tumors that have spread from where they started to nearby tissue or lymph nodes (locally advanced) or have spread from the primary site (place where they started) to other places in the body (metastatic). Nintedanib may stop the growth of tumor cells by slowing or stopping a certain type of receptor called vascular endothelial growth factor receptor (VEGFR) from attaching to its target. This may stop the growth of neuroendocrine tumors by blocking the growth of new blood vessels necessary for tumor growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess progression free survival (PFS), defined as the time interval from initiation of therapy, to its cessation for documentation of progressive disease (PD) or death.

SECONDARY OBJECTIVES:

I. To assess the clinical response (complete response + partial response) in all patients with measurable disease (using standard Response Evaluation Criteria in Solid Tumors [RECIST] version [v]1.1 criteria).

II. To assess overall survival (OS) in all patients. III. Assess changes in quality of life (QOL) throughout treatment using the European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) - Gastrointestinal Neuroendocrine Tumors (NET) 21 (GI.NET21) questionnaire for carcinoid patients with gastrointestinal neuroendocrine tumors, in all patients who have filled out at least two QOL questionnaires and, will be reported by groups based on response (response, stable disease or progressive disease).

IV. Steady-state pharmacokinetics (PK) of nintedanib, biomarkers, regulatory T cell (Treg) and cytokine expression and growth factors will be analyzed for all patients and reported in groups based on response.

V. Gene mutations and copy number alterations analysis in the mammalian target of rapamycin (mTOR) pathway (will be performed only on the first 10 patients), protein expression of activation of protein kinase B (Akt) (as well as other downstream targets).

VI. Toxicity (graded using the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version 4.0) will be closely monitored and all toxicities will be tabulated.

OUTLINE:

Patients receive nintedanib orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be on a stable dose of octreotide (Sandostatin®) long-acting release (LAR) or lanreotide for 3 months prior to study enrollment
* Patient must have histologically or cytologically confirmed well differentiated or moderately differentiated (low grade or intermediate grade) neuroendocrine tumor that is locally advanced or metastatic and not of pancreatic origin
* Measurable disease determined by computed tomography (CT) or magnetic resonance imaging (MRI)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Life expectancy greater than 3 months
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Total bilirubin =< 2 mg/dL
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 1.5 x upper limit of normal (ULN) and bilirubin =< ULN for patients without liver metastases
* AST/ALT =< 2.5 x ULN and bilirubin =< ULN for patients with liver metastases
* Patients with Gilbert syndrome and bilirubin < 2 x ULN and normal AST/ALT
* Creatinine =< 1.5 mg/dl
* Prior treatment will be permitted including surgery (>= 4 weeks), cytotoxic chemotherapy (maximum of 2 prior regimens); radiation, interferon, targeted growth factors (>= 4 weeks); and prior treatment with octreotide, will be allowed
* Ability to swallow and retain oral medication
* Participants of child-bearing potential (both male and female) must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Archival tissue of carcinoid biopsy must be available

Exclusion Criteria:

* Uncontrolled hypertension, unstable angina, New York Heart Association grade II or greater congestive heart failure, unstable symptomatic arrhythmia requiring medication, or clinically significant peripheral vascular disease (grade II or greater)
* Presence of brain metastases
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 0, or anticipated need for major surgical procedure during the course of the study, or fine needle aspirations or core biopsies within 7 days prior to day 0
* Significant proteinuria at baseline (>= 500 mg/24 hours [h])
* Serious non-healing wound, ulcer or bone fracture
* Evidence of bleeding diathesis or coagulopathy
* Recent (=< 6 months) arterial thromboembolic events, including transient ischemic attack, cerebrovascular accident, unstable angina, or myocardial infarction
* Poorly differentiated neuroendocrine carcinoma, high-grade neuroendocrine carcinoma, adenocarcinoid, goblet cell carcinoma, or small cell carcinoma
* Hepatic artery embolization or ablation of hepatic metastasis within 3 months of enrollment, prior peptide receptor radionuclide therapy (PRRT) within 4 months or any other cancer therapy within 4 weeks (as long as all toxicities are resolved)
* Intolerance or hypersensitivity to octreotide
* Severe or uncontrolled medical conditions
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renuka Iyer, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Nintedanib)
Started | 32
Completed | 30
Not Completed | 2
Not completed — bowel obstruction (unrelated to dis-ease) | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 16
Age, Continuous [Median (Full Range); unit: years] | 65 [45 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: PFS
Description: Will be reported using standard Kaplan-Meier methods. Ninety percent confidence intervals for the median PFS will be calculated using Greenwood's formula. Additionally, a confidence interval for the 16-week PFS rate will be obtained using Jeffrey's prior method. The association between survival and quantified variables will be investigated using the Cox-proportional hazard model.
Time Frame: Time interval from initiation of therapy, to its cessation for documentation of PD or death, assessed up to 2 years
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 30
months | 11 [5.5 to 19.3]

2. Secondary Outcome: Change in Quality of Life Score
Description: Quality of life will be investigated calculated by Subjects filing out EORTC Gastrointestinal Neuroendocrine Tumour 21 Questionnaire (QLQ-GI.NET21) A 21 question questionnaire that use a 4-point scale (1 = Not at all, 2 = A little, 3 = Quite a bit, 4 = Very much). The scores for different scales (i.e. endocrine, gastrointestinal, treatment, social function, disease Related, and global) are calculated by summing related questions from the questionnaire. The range of the subscale scores are from 0 to 100, with higher scores being worse.
  After the subscale scores being calculated, the Change in quality of life is calculated by subtracting baseline score from end of treatment
Time Frame: Baseline to 30 days post-treatment
Population: Patients completed at least 2 EORTC QLQ-GI.NET21 questionnaires are included for this outcome estimate
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 31
score on a scale
  Change in endocrine scale | 0 [-44 to 33]
  Change in gastrointestinal scale | 0 [-3 to 5]
  Change in treatment scale | 0 [-50 to 44]
  Change in social function scale | 0 [-44 to 33]
  Change in Disease Related Worry Scale | -6 [-67 to 56]
  Change in Global scale | 1 [-21 to 31]

3. Secondary Outcome: Plasma Concentrations at Steady State (Cpre,ss) of Nintedanib at Baseline and Week 8
Description: Sample collection will be obtained at baseline and week 8
Time Frame: Baseline to week 8
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 32
ng/mL | 11.2 [0.9 to 171.0]

4. Secondary Outcome: Clinical Response (Complete Response + Partial Response) Measured Using Standard RECISTv1.1 Criteria
Description: Exact 90% confidence interval estimates using the Clopper-Pearson method will be given for the response rates. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI, response rates are categorized as Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 28
Participants
  SD | 26
  PD | 1
  PR | 1

5. Secondary Outcome: Median OS
Description: Will be reported using standard Kaplan-Meier methods. Ninety-five percent confidence intervals for the median OS will be calculated using Greenwood's formula. The association between survival and quantified variables will be investigated using the Cox-proportional hazard model.
Time Frame: Up to 3 years (telephone contact is acceptable).
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 32
months | 32.7 [27.6 to NA] — 90% Upper Confidence Interval was not reached (Not Available), because not enough people deceased to estimate the upper confidence

6. Secondary Outcome: Ratio of FGFR IIIb/IIIc and Ki-67 and Microvessel Density Scores
Description: Scores will be obtained to investigate association with PFS, clinical response, QOL and survival.
Time Frame: Baseline
Population: The FGFR IIIb/IIIcm, Ki-67m and microvessel density scores were not measured (i.e. data not obtained) and analyses were not performed.
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Biomarker Levels
Description: Will be analyzed for all patients and reported in groups based on response.
Time Frame: Baseline
Population: The appropriate biomarkers were not measured (i.e. data not obtained) and analyses were not performed.
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Change in Cytokine Expression
Description: Will be analyzed for all patients and reported in groups based on response. Changes in pre- and post-treatment cytokine expression will be analyzed using permutation paired t-tests.
Time Frame: Baseline to 8 weeks
Population: The appropriate cytokine expressions were not measured (i.e. data not obtained) and analyses were not performed.
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Change in Growth Factors
Description: Will be analyzed for all patients and reported in groups based on response. Changes in pre- and post-treatment growth factors will be analyzed using permutation paired t-tests.
Time Frame: Baseline to 30 days post-treatment
Population: The appropriate growth factors were not measured (i.e. data not obtained) and analyses were not performed.
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Gene Mutations and Copy Number Alterations
Description: Gene mutations and copy number alterations in the several pathways particularly mTOR pathway will be evaluated. Will be analyzed for all patients and correlated with clinical outcomes.
Time Frame: Baseline
Population: Gene mutations and copy number alterations were not measured (i.e. data not obtained) and analyses were not performed.
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Treg Levels
Description: Will be analyzed for all patients and reported in groups based on response.
Time Frame: Baseline
Population: Treg levels were not measured and analyses were not performed.
Arm/Group | Treatment (Nintedanib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Routine AEs occurring at baseline, Cycle 1-Week 1-Day 1, Cycle 1-Week 3-Day 1, Day 1 of subsequent cycles, End of Treatment, and PFS Follow-Up, will be reported, up to 33 months.
Arm/Group | Treatment (Nintedanib)
All-Cause Mortality (participants affected / at risk) | 18/32
Serious Adverse Events (participants affected / at risk) | 14/32
Other Adverse Events (participants affected / at risk) | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nintedanib) (N=32)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (3)
Myocardial infarction (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Early satiety (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Therapeutic response decreased (General disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nintedanib) (N=32)
Anaemia (Blood and lymphatic system disorders) | 9 (13)
Leukocytosis (Blood and lymphatic system disorders) | 3 (4)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Aortic valve disease (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Tricuspid valve disease (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Eye disorder (Eye disorders) | 1 (1)
Photopsia (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 10 (20)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1)
Angular cheilitis (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 12 (19)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Faeces pale (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 19 (28)
Oral dysaesthesia (Gastrointestinal disorders) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Tooth discolouration (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 12 (17)
Chills (General disorders) | 2 (2)
Fatigue (General disorders) | 12 (20)
Influenza like illness (General disorders) | 5 (5)
Infusion site extravasation (General disorders) | 1 (1)
Localised oedema (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (3)
Oedema peripheral (General disorders) | 4 (5)
Peripheral swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Contrast media allergy (Immune system disorders) | 1 (1)
Cellulitis (Infections and infestations) | 2 (3)
Gastroenteritis (Infections and infestations) | 1 (1)
Hepatic infection (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (2)
Peritonitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (2)
Stoma site infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 7 (7)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (4)
Stoma site pain (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 9 (16)
Aspartate aminotransferase increased (Investigations) | 11 (27)
Bacterial test positive (Investigations) | 1 (1)
Blood alkaline phosphatase (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 11 (19)
Blood bilirubin increased (Investigations) | 5 (11)
Blood creatine increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 3 (4)
Blood glucose increased (Investigations) | 1 (1)
Brain natriuretic peptide (Investigations) | 1 (1)
Haemoglobin increased (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 2 (4)
Lymphocyte count decreased (Investigations) | 16 (57)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 12 (16)
Troponin I increased (Investigations) | 3 (3)
Weight decreased (Investigations) | 13 (19)
Weight increased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 9 (21)
White blood cell count increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 8 (10)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 16 (46)
Hypernatraemia (Metabolism and nutrition disorders) | 3 (8)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 (18)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (9)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (6)
Dysgeusia (Nervous system disorders) | 6 (8)
Headache (Nervous system disorders) | 6 (7)
Memory impairment (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (4)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Stress (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (5)
Chronic kidney disease (Renal and urinary disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1)
Nipple pain (Reproductive system and breast disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (2)
Hair colour changes (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Edentulous (Social circumstances) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1)
Flushing (Vascular disorders) | 5 (5)
Hypertension (Vascular disorders) | 17 (38)
Hypotension (Vascular disorders) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT02399215/Prot_SAP_000.pdf